CLINICAL TRIAL: NCT03704155
Title: Effect of Botulinum Toxin Type A Associated With Physical Therapy on the Functional Capacity of Children With Spastic Cerebral Palsy: A Randomized Controlled Clinical Trial
Brief Title: Effect of Botulinum Toxin Type A Associated With Physical Therapy on Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Claudia Santos Oliveira (Unknown); Daniela Aparecida Biasotto-Gonzalez (Unknown)
Responsible Party: Principal Investigator, Fabiano Politti, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTA
Record Dates: First submitted 2018-07-04; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy, Spastic; Physical Therapy; Botulinum Toxin
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Evaluator 1: triage, random draw of treatments to be performed; Evaluator 2: BoNT-A application; Evaluator 3: assessment data collection; Evaluator 4: physical therapy treatment. Evaluator 3 was blinded in relation to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (EG) (Experimental): The EG was treated with Botulinum toxin type A and physiotherapy (stretching, balancing training, functional walking training).
  Interventions: Drug: Botulinum toxin type A; Other: Physical Therapy
- Control group (CG) (Active Comparator): GC was treated with physiotherapy (stretching, balancing training, functional walking training).
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum Toxin type A The intervention with BoNT-A (Dysport®, Ipsen Biopharmaceutical, USA) was performed in the gastrocnemius and soleus muscles, bilaterally for diplegic children and unilaterally for hemiplegic children.
  Arms: Experimental group (EG)
Other: Physical Therapy — Physiotherapeutic intervention was performed twice a week, with duration of one hour per session for 4 weeks. To maintain standardization of treatment, physiotherapists received a booklet with instructions on what treatment they should do.
  The intervention protocol consisted of:
  * Passive stretching of lower limbs,
  * Stretching associated with the functionality of the plantar flexor muscles, knee flexors, adductors and hip flexors;
  * Strengthening of the antagonist muscles with the application of BoNT-A;
  * Static and dynamic balance training;
  * Up and down stairs;
  * Functional walking training, prioritizing the initial contact of the heel and active and passive dorsiflexion.

SUMMARY:
Purpose: The aim of this study was investigate the effects of botulinum toxin type A (BoNT-A) associated with physical therapy on the functional capacity of children with spastic cerebral palsy (CP). Material and methods: Twenty-four children with spastic CP were concealed and randomly assigned to the Experimental Group (EG) consisting of 12 patients treated with BoNT-A and physical therapy and Control with 12 patients treated only with physical therapy. All participants were assessed through motor and functional scales (GMFM-88, Ashworth, Berg Balance Scale, TUG test and Pediatric Evaluation of Disability Inventory) at three different times: before and after 30 days of treatment as well as 3 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spastic Cerebral Palsy
* Clinical diagnosis of Dynamic equine feet

Exclusion Criteria:

* Use of phenol in the last 12 months
* Neurological blocks in the last 6 months
* Clinical diagnosis of structured orthopedic deformities with surgical indications

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Severity of muscle hypertonia | 3 months
  The classification of hypertonia was performed by Modified Ashworth Scale
Functional balance | 3 months
  Functional balance was assessed using the Berg Balance Scale (BBS).

SECONDARY OUTCOMES:
Functional mobility | 3 months
  Functional mobility was performed by The Timed Up and Go test (TUG test).
Functional performance | 3 months
  Functional performance was assessed using Pediatric Evaluation of Disability Inventory (PEDI).

IPD SHARING:
Plan to Share IPD: No